CLINICAL TRIAL: NCT04488952
Title: The Effects of Different Anesthesia Methods on Perioperative Neurocognitive Disorders in the Elderly: a Randomized Controlled Trial
Brief Title: The Effects of Different Anesthesia Methods on Perioperative Neurocognitive Disorders in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, ZhiHeng Liu, Chair of Department of Anesthesiology, Shenzhen Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20193357001-XZ01
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: PND
Keywords: PND,anesthesia method, elderly
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nerve block combined with general anesthesia group (Experimental): Patients in this group receive nerve block combined with general anesthesia.
  Interventions: Device: nerve block combined with general anesthesia; Device: spinal anesthesia
- spinal anesthesia group (Experimental): Patients in this group receive spinal anesthesia.
  Interventions: Device: nerve block combined with general anesthesia; Device: spinal anesthesia
- control group (Placebo Comparator): This group is used to obtain the learning effect.
  Interventions: Device: nerve block combined with general anesthesia; Device: spinal anesthesia

INTERVENTIONS:
Device: nerve block combined with general anesthesia — Patients in this group receive nerve block combined with general anesthesia.
Device: spinal anesthesia — Patients in this group receive spinal anesthesia.

SUMMARY:
Perioperative Neurocognitive Disorders(PND) is a common perioperative complication among the elderly, especially in the plastic surgery. Different anesthesia methods have different incidences of PND, but it's still unknow which is better between spinal anesthesia and nerve block combined with general anesthesia. We will apply a psychometric battery test which contain different cognitive domains to estimate the incidence of PND at a week a month and a year after surgery with different anesthesia methods. Study has showed that functional magnetic resonance imaging (fMRI) could detect a cognitive decline through spontaneous neuronal activity in the cortex and hippocampus. In our study, multi-mode imaging technology is used to conduct in-depth research on MRI and make correlation analysis with cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-85years
* ASA I-III
* Received elective surgery of unilateral lower extremity orthopedics
* The anesthesia lasted more than 2 hours

Exclusion Criteria:

-

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PND seven days after surgery | seven days after surgery

SECONDARY OUTCOMES:
Incidence of PND one month after surgery | one month after surgery
Incidence of PND one year after surgery | one year after surgery
Hospital stay | one to two weeks after surgery
Number of patients entrance the ward of ICU after surgery | one week post-operation
Mortality rate | one year after surgery
Postoperative complications | one month post-operation
ADL of frontal lobe，temporal lobe and occipital lobe | one day pre-operation, one week post-operation
ADL of frontal lobe | one day pre-operation, one week post-operation
BOLD of the whole brain | one day pre-operation, one week post-operation
ADL of temporal lobe | one day pre-operation, one week post-operation
ADL of occipital lobe | one day pre-operation, one week post-operation
One year event-free survival | one year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bittner EA, Yue Y, Xie Z. Brief review: anesthetic neurotoxicity in the elderly, cognitive dysfunction and Alzheimer's disease. Can J Anaesth. 2011 Feb;58(2):216-23. doi: 10.1007/s12630-010-9418-x. Epub 2010 Dec 21. PMID 21174183
- [Background] Yildizeli B, Ozyurtkan MO, Batirel HF, Kuscu K, Bekiroglu N, Yuksel M. Factors associated with postoperative delirium after thoracic surgery. Ann Thorac Surg. 2005 Mar;79(3):1004-9. doi: 10.1016/j.athoracsur.2004.06.022. PMID 15734423
- [Background] Mason SE, Noel-Storr A, Ritchie CW. The impact of general and regional anesthesia on the incidence of post-operative cognitive dysfunction and post-operative delirium: a systematic review with meta-analysis. J Alzheimers Dis. 2010;22 Suppl 3:67-79. doi: 10.3233/JAD-2010-101086. PMID 20858956
- [Background] Alkire MT, Pomfrett CJ, Haier RJ, Gianzero MV, Chan CM, Jacobsen BP, Fallon JH. Functional brain imaging during anesthesia in humans: effects of halothane on global and regional cerebral glucose metabolism. Anesthesiology. 1999 Mar;90(3):701-9. doi: 10.1097/00000542-199903000-00011. PMID 10078670
- [Background] Peng L, Xu L, Ouyang W. Role of peripheral inflammatory markers in postoperative cognitive dysfunction (POCD): a meta-analysis. PLoS One. 2013 Nov 13;8(11):e79624. doi: 10.1371/journal.pone.0079624. eCollection 2013. PMID 24236147
- [Background] Silbert B, Evered L, Scott DA, McMahon S, Choong P, Ames D, Maruff P, Jamrozik K. Preexisting cognitive impairment is associated with postoperative cognitive dysfunction after hip joint replacement surgery. Anesthesiology. 2015 Jun;122(6):1224-34. doi: 10.1097/ALN.0000000000000671. PMID 25859906
- [Background] Squire LR. Memory and the hippocampus: a synthesis from findings with rats, monkeys, and humans. Psychol Rev. 1992 Apr;99(2):195-231. doi: 10.1037/0033-295x.99.2.195. PMID 1594723
- [Background] Zola-Morgan S, Squire LR, Amaral DG. Human amnesia and the medial temporal region: enduring memory impairment following a bilateral lesion limited to field CA1 of the hippocampus. J Neurosci. 1986 Oct;6(10):2950-67. doi: 10.1523/JNEUROSCI.06-10-02950.1986. PMID 3760943
- [Background] Price CC, Tanner JJ, Schmalfuss I, Garvan CW, Gearen P, Dickey D, Heilman K, McDonagh DL, Libon DJ, Leonard C, Bowers D, Monk TG. A pilot study evaluating presurgery neuroanatomical biomarkers for postoperative cognitive decline after total knee arthroplasty in older adults. Anesthesiology. 2014 Mar;120(3):601-13. doi: 10.1097/ALN.0000000000000080. PMID 24534857
- [Background] Hole A, Terjesen T, Breivik H. Epidural versus general anaesthesia for total hip arthroplasty in elderly patients. Acta Anaesthesiol Scand. 1980 Aug;24(4):279-87. doi: 10.1111/j.1399-6576.1980.tb01549.x. PMID 7468115
- [Background] Berggren D, Gustafson Y, Eriksson B, Bucht G, Hansson LI, Reiz S, Winblad B. Postoperative confusion after anesthesia in elderly patients with femoral neck fractures. Anesth Analg. 1987 Jun;66(6):497-504. PMID 3578861
- [Background] Williams-Russo P, Sharrock NE, Mattis S, Szatrowski TP, Charlson ME. Cognitive effects after epidural vs general anesthesia in older adults. A randomized trial. JAMA. 1995 Jul 5;274(1):44-50. PMID 7791257
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] O'Hara DA, Duff A, Berlin JA, Poses RM, Lawrence VA, Huber EC, Noveck H, Strom BL, Carson JL. The effect of anesthetic technique on postoperative outcomes in hip fracture repair. Anesthesiology. 2000 Apr;92(4):947-57. doi: 10.1097/00000542-200004000-00011. PMID 10754613
- [Background] Chen MH, Liao Y, Rong PF, Hu R, Lin GX, Ouyang W. Hippocampal volume reduction in elderly patients at risk for postoperative cognitive dysfunction. J Anesth. 2013 Aug;27(4):487-92. doi: 10.1007/s00540-012-1548-6. Epub 2013 Jan 31. PMID 23371369
- [Background] Maekawa K, Baba T, Otomo S, Morishita S, Tamura N. Low pre-existing gray matter volume in the medial temporal lobe and white matter lesions are associated with postoperative cognitive dysfunction after cardiac surgery. PLoS One. 2014 Jan 27;9(1):e87375. doi: 10.1371/journal.pone.0087375. eCollection 2014. PMID 24475280
- [Background] Wei M, Shi J, Li T, Ni J, Zhang X, Li Y, Kang S, Ma F, Xie H, Qin B, Fan D, Zhang L, Wang Y, Tian J. Diagnostic Accuracy of the Chinese Version of the Trail-Making Test for Screening Cognitive Impairment. J Am Geriatr Soc. 2018 Jan;66(1):92-99. doi: 10.1111/jgs.15135. Epub 2017 Nov 14. PMID 29135021
- [Background] Ruff RM, Light RH, Parker SB, Levin HS. The psychological construct of word fluency. Brain Lang. 1997 May;57(3):394-405. doi: 10.1006/brln.1997.1755. PMID 9126423
- [Background] Shi J, Tian J, Wei M, Miao Y, Wang Y. The utility of the Hopkins Verbal Learning Test (Chinese version) for screening dementia and mild cognitive impairment in a Chinese population. BMC Neurol. 2012 Nov 7;12:136. doi: 10.1186/1471-2377-12-136. PMID 23130844
- [Background] Norkiene I, Samalavicius R, Ivaskevicius J, Budrys V, Paulauskiene K. Asymptomatic carotid artery stenosis and cognitive outcomes after coronary artery bypass grafting. Scand Cardiovasc J. 2011 Jun;45(3):169-73. doi: 10.3109/14017431.2011.562525. Epub 2011 Mar 15. PMID 21405959
- [Background] Knopman DS, Roberts RO, Geda YE, Pankratz VS, Christianson TJ, Petersen RC, Rocca WA. Validation of the telephone interview for cognitive status-modified in subjects with normal cognition, mild cognitive impairment, or dementia. Neuroepidemiology. 2010;34(1):34-42. doi: 10.1159/000255464. Epub 2009 Nov 5. PMID 19893327
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Background] Li WX, Luo RY, Chen C, Li X, Ao JS, Liu Y, Yin YQ. Effects of propofol, dexmedetomidine, and midazolam on postoperative cognitive dysfunction in elderly patients: a randomized controlled preliminary trial. Chin Med J (Engl). 2019 Feb;132(4):437-445. doi: 10.1097/CM9.0000000000000098. PMID 30707179